CLINICAL TRIAL: NCT00792818
Title: The Efficacy and Safety of Curcuma Domestica Extracts and Ibuprofen for Therapy of Patients With Knee Osteoarthritis, the Randomized Double-blinded Controlled Trial, Multicenter Study
Brief Title: The Efficacy and Safety of Curcuma Domestica Extracts and Ibuprofen in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Vilai Kuptniratsaikul, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si134/2008
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Knee, Curcumin, Multicenter, RCT
MeSH Terms: conditions — Osteoarthritis | interventions — Curcumin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcuma domestica (Experimental): 1,500 mg/day (oral) divided into 3 times for 28 days
  Interventions: Drug: Curcuma domestica extracts
- Ibuprofen (Active Comparator): 1,200 mg/day (oral) divided into 3 times for 28 days
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Curcuma domestica extracts — 1,500 mg per day (oral)divided into 3 times for 28 days
  Other Names: Curcumin
  Arms: curcuma domestica
Drug: Ibuprofen — 1,200 mg/days (oral) divided into 3 times for 28 days
  Other Names: Brufen
  Arms: Ibuprofen

SUMMARY:
Osteoarthritis of knee is common degenerative musculoskeletal diseases. Non-steroidal antiinflammatory drugs (NSAIDs) are used to decrease pain symptom but someone can not tolerate its gastrointestinal adverse effects. In vitro studies showed that curcumin had an inhibitory effect on substances playing an important role in inflammatory pathway. The mechanisms by which curcumin prevents inflammation are postulated through inhibition of many cytokines, for example, lipo-oxygenase, cyclo-oxygenase, and phospholipase. Therefore, if curcumin is effective as NSAIDs with less side effects, it can be an alternative treatment for those OA knee patients.

DETAILED DESCRIPTION:
Curcumin was demonstrated to be safe and had anti-inflammatory activity in six studies in humans. It may exert its anti-inflammatory activity by inhibition of a number of different molecules that play a role in inflammation.

Our experience in a study of 100 subjects revealed a trend towards a greater effect in OA patients receiving Curcuma domestica extracts. However, studies with adequate sample and dosage of Ibuprofen are recommended to demonstrate the efficacy of C.domestica extracts in alleviating knee pain and improving knee functions.

The objective of the study was to determine the efficacy and safety of C.domestica extracts in pain reduction and functional improvement in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis
* Knee pain score more than or equal to 5 point (NRS 0-10)
* Age >= 50 years, not > 75 years
* Knee crepitus
* Knee stiffness less than 30 minutes
* Urine pregnancy test negative in case of not being menopausal period

Exclusion Criteria:

* History of GI ulcer or melena
* Having hepatic or bile duct diseases(SGOT ≥ 37 u/L, SGPT ≥ 40 u/L)
* Having renal disease or abnormal renal functions (serum creatinine ≥ 1.5 mg/dl)
* Asthma or gout
* Allergy to ibuprofen or curcumin
* History of intraarticular knee injection within 6 months
* Post knee arthroplasty
* History of intermittent claudication
* Unable to walk, for example hemiplegia, severe lung/heart diseases
* Knee x-ray found chondrocalcinosis
* On anticoagulant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in mean WOMAC pain subscale | 12 months

SECONDARY OUTCOMES:
Adverse events | 12 months
Quality of life: SF-36 | 12 months
Change in WOMAC score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vilai - Kuptniratsaikul, MD., Principal Investigator — Mahidol University
Locations (6):
- Thailand (6):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - KhonKaen University Hospital, KhonKaen
  - VachiraPhuket Hospital, Phuket
  - Rajburi Hospital, Ratchaburi
  - Songkla Hospital, Songkhla

REFERENCES:
- [Derived] Kuptniratsaikul V, Dajpratham P, Taechaarpornkul W, Buntragulpoontawee M, Lukkanapichonchut P, Chootip C, Saengsuwan J, Tantayakom K, Laongpech S. Efficacy and safety of Curcuma domestica extracts compared with ibuprofen in patients with knee osteoarthritis: a multicenter study. Clin Interv Aging. 2014 Mar 20;9:451-8. doi: 10.2147/CIA.S58535. eCollection 2014. PMID 24672232